CLINICAL TRIAL: NCT02878603
Title: Prospective Follow-up Study for Patients Who Completed Study ALX0681-C301 (HERCULES) to Evaluate Long-term Safety and Efficacy of Caplacizumab (Post-HERCULES)
Brief Title: Follow-up Study for Patients Who Completed Study ALX0681-C301 (Post-HERCULES)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTS16371; 2016-001503-23 (EudraCT Number); ALX0681-C302 (Other: Ablynx)
Record Dates: First submitted 2016-08-04; First posted 2016-08-25 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Acquired Thrombotic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombotic Thrombocytopenic | interventions — caplacizumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- caplacizumab (Experimental): Participants who completed study ALX0681-C301 (NCT02553317) with standard of care (plasma exchange [PE], corticosteroid and other immunosuppressive agents) or caplacizumab with PE and immunosuppressive agents were enrolled in study LTS16371. Participants upon each recurrence of aTTP in LTS16371 and not meeting any criteria (namely: pregnancy, history of severe and/or serious hypersensitivity reaction to investigational medicinal product [IMP], withdrawal before receiving IMP, received more than 1 PE) were treated with caplacizumab initial 10 milligrams (mg) intravenous dose followed by a daily 10 mg subcutaneous injections during the period of PE and for 30 days after stop of PE (and eventually 28-day extension period, if needed). Participants with or without recurrence were followed up twice yearly up to maximum of 36 months in LTS16371.
  Interventions: Biological: Caplacizumab; Other: Standard of Care

INTERVENTIONS:
Biological: Caplacizumab
Other: Standard of Care — • PE with plasma (e.g., fresh frozen plasma, solvent detergent/viral-inactivated plasma, cryosupernatant), • Corticosteroid treatment and • Use of other immunosuppressive agents (e.g., rituximab).

SUMMARY:
The objectives of this study were to evaluate long-term safety and efficacy of caplacizumab, to evaluate safety and efficacy of repeated use of caplacizumab and to characterize long-term impact of acquired thrombotic thrombocytopenic purpura (aTTP).

ELIGIBILITY:
Inclusion Criteria:

1. Completed the Final (28 day) follow-up visit in Study ALX0681-C301.
2. >= 18 years of age at the time of signing the informed consent form.
3. Provided informed consent prior to initiation of any study specific activity/procedure.

Exclusion Criteria:

1. Not being able/willing to comply with the study protocol procedures.
2. Currently enrolled in a clinical study with another investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2020-10-23 (Actual); Study Completion 2020-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Ablynx, MD, Study Director — Ablynx NV
Locations (45):
- United States (8):
  - Investigator site, St Louis, Missouri
  - Investigator site, Valhalla, New York
  - Investigator Site, Durham, North Carolina
  - Investigator Site, Columbus, Ohio
  - Investigator Site, Oklahoma City, Oklahoma
  - Investigator site, Pittsburgh, Pennsylvania
  - Investigator Site, Charleston, South Carolina
  - Investigator site, Greenville, South Carolina
- Investigator site, Vienna, Austria
- Belgium (4):
  - Investigator site, Antwerp
  - Investigator site, Brussels
  - Investigator site, La Louvière
  - Investigator site, Leuven
- Canada (3):
  - Investigator Site, Halifax
  - Investigator Site, Québec
  - Investigator Site, Toronto
- Czechia (2):
  - Investigator Site, Brno
  - Investigator Site, Olomouc
- France (5):
  - Investigator site, Caen
  - Investigator site, Lille
  - Investigator site, Marseille
  - Investigator site 1, Paris
  - Investigator site 2, Paris
- Hungary (2):
  - Investigator Site, Budapest
  - Investigator Site, Debrecen
- Israel (3):
  - Investigator Site, Haifa
  - Investigator Site, Jerusalem Region
  - Investigator Site, Nahariya
- Italy (5):
  - Investigator Site, Catania
  - Investigator Site, Milan
  - Investigator site, Pesaro
  - Investigator Site, Rome
  - Investigator Site, Vicenza
- Spain (5):
  - Investigator Site 1, Barcelona
  - Investigator Site 2, Barcelona
  - Investigator site, Seville
  - Investigator Site 2, Valencia
  - Investyigator Site 1, Valencia
- Investigator site, Bern, Switzerland
- Turkey (Türkiye) (3):
  - Investigator site, Ankara
  - Investigator site, Istanbul
  - Investigator site, Kayseri
- United Kingdom (3):
  - Investigator Site, Bristol
  - Investigator site, Liverpool
  - Investigator Site, London

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Scully M, de la Rubia J, Pavenski K, Metjian A, Knobl P, Peyvandi F, Cataland S, Coppo P, Kremer Hovinga JA, Minkue Mi Edou J, De Passos Sousa R, Callewaert F, Gunawardena S, Lin J. Long-term follow-up of patients treated with caplacizumab and safety and efficacy of repeat caplacizumab use: Post-HERCULES study. J Thromb Haemost. 2022 Dec;20(12):2810-2822. doi: 10.1111/jth.15892. Epub 2022 Oct 21. PMID 36138517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 43 active sites in 13 countries. A total of 104 participants who completed Study ALX0681-C301 (HERCULES; NCT02553317) were enrolled between 06-October-2016 and 27-October-2017 in this current study: LTS16371 (ALX0681-C302).
Pre-assignment Details: Participants who were randomized to caplacizumab/placebo and received caplacizumab for recurrence of acquired thrombotic thrombocytopenic purpura (aTTP) in ALX0681-C301 were enrolled in Caplacizumab group, and participants randomized to placebo in ALX0681-C301 were enrolled under Standard of Care (SoC) group in the current study LTS16371.
Groups:
- Standard of Care (SoC) (Treated in Study C301): Participants who completed study ALX0681-C301 with SoC (plasma exchange [PE], corticosteroid and other immunosuppressive agents) treatment were enrolled in study LTS16371. Participants upon each recurrence of aTTP in LTS16371 and not meeting any criteria (namely: pregnancy, history of severe and/or serious hypersensitivity reaction to investigational medicinal product [IMP], withdrawal before receiving IMP, received more than 1 PE) were treated with caplacizumab initial 10 mg intravenous (IV) dose followed by a daily 10 milligrams (mg) subcutaneous (SC) injections during the period of PE and for 30 days after stop of PE (and eventually 28-day extension period, if needed). Participants with or without recurrence were followed up twice yearly up to maximum of 36 months in LTS16371.
- Caplacizumab (Treated in Study C301): Participants who completed study ALX0681-C301 and received caplacizumab with PE and immunosuppressive agents were enrolled in study LTS16371. Participants upon each recurrence of aTTP in LTS16371 and not meeting any criteria (namely: pregnancy, history of severe and/or serious hypersensitivity reaction to IMP, withdrawal before receiving IMP, received more than 1 PE) were treated with caplacizumab initial 10 mg IV dose followed by a daily 10 mg SC injections during the period of PE and for 30 days after stop of PE (and eventually 28-day extension period, if needed). Participants with or without recurrence were followed up twice yearly up to maximum of 36 months in LTS16371.
Period: Overall Study
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Started | 29 | 75
Completed | 23 | 70
Not Completed | 6 | 5
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Death | 1 | 0
Not completed — Physician Decision | 0 | 3

BASELINE CHARACTERISTICS:
Population: Analyzed on overall intention-to-observe (overall ITO) population which included participants who were enrolled in LTS16371, grouped by whether they received caplacizumab during previous study ALX0681-C301 versus those who never received caplacizumab before enrollment in LTS16371.
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301) | Total Title
Number analyzed (Participants) | 29 | 75 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (14.8) | 46.0 (11.9) | 47.5 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 51 | 74
  Male | 6 | 24 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 13 | 19
  White | 21 | 52 | 73
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Acquired Thrombotic Thrombocytopenic Purpura (aTTP) Related Events
Description: aTTP-related events were defined as: aTTP-related death, recurrence of aTTP (defined as recurrent thrombocytopenia requiring initiation of daily PE) or at least one major thromboembolic event (e.g., myocardial infarction, cerebrovascular accident, pulmonary embolism, or deep venous thrombosis). Percentage of participants with at least one aTTP-related events during the study were reported in this outcome measure.
Time Frame: From Baseline up to 36 months
Population: Analysis was performed on efficacy intention-to-observe (efficacy ITO) population which included participants who were enrolled in LTS16371 and did not experience an aTTP recurrence in previous study ALX0681-C301 or prior to the beginning of LTS16371.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
percentage of participants | 37.9 | 8.2

2. Primary Outcome: Number of Acquired Thrombotic Thrombocytopenic Purpura-related Events
Description: aTTP-related events were defined as: aTTP-related death, recurrence of aTTP (defined as recurrent thrombocytopenia requiring initiation of daily PE) or at least one major thromboembolic event (e.g., myocardial infarction, cerebrovascular accident, pulmonary embolism or deep venous thrombosis).
Time Frame: From Baseline up to 36 months
Population: Analysis was performed on efficacy ITO population which included participants who were enrolled in LTS16371 and did not experience an aTTP recurrence in previous study ALX0681-C301 or prior to the beginning of LTS16371.
Measure: Number; unit: aTTP-related events
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
aTTP-related events | 11 | 4

3. Primary Outcome: Time to First Acquired Thrombotic Thrombocytopenic Purpura-related Events
Description: Time to first aTTP-related events was defined as the duration of time (in days) from Baseline up to first aTTP-related event in LTS16371. Participants without an event during LTS16371 were censored at the end of the study. Kaplan-Meier method was used for the analysis.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
days | NA [845.00 to NA] — Median and upper limit of 95% confidence interval (CI) were not calculated due to very few participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not calculated due to very few participants with events.

4. Primary Outcome: Number of Participants With aTTP Related Deaths Reported During the Study
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
Participants | 1 | 0

5. Primary Outcome: Percentage of Participants With Recurrence of Disease (aTTP)
Description: Recurrence of aTTP was defined as recurrent thrombocytopenia requiring initiation of daily PE.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
percentage of participants | 27.6 | 8.2

6. Primary Outcome: Number of Disease (aTTP) Recurrence Reported During the Study
Description: Recurrence of aTTP was defined as recurrent thrombocytopenia requiring initiation of daily PE.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Number; unit: aTTP recurrences
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
aTTP recurrences | 8 | 4

7. Primary Outcome: Time to Recurrence of Disease (aTTP)
Description: Time to first recurrence of disease (aTTP) was defined as the duration of time (in days) from Baseline up to first recurrence of aTTP event in LTS16371. Recurrence of aTTP: defined as recurrent thrombocytopenia requiring initiation of daily PE. Participants without an event during LTS16371 were censored at the end of the study. Kaplan-Meier method was used for the analysis.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
days | NA [1280.00 to NA] — Median and upper limit of 95% CI were not calculated due to very few participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not calculated due to very few participants with events.

8. Primary Outcome: Percentage of Participants With Major Thromboembolic Events Including Thrombotic Thrombocytopenic Purpura (TTP)
Description: Major thromboembolic events (e.g., myocardial infarction, cerebrovascular accident, pulmonary embolism, or deep venous thrombosis) were assessed based on Standardized Medical Dictionary for Regulatory Activities (MedDRA) Query (SMQ). Reported major thromboembolic events included TTP recurrences.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
percentage of participants | 37.9 | 8.2

9. Primary Outcome: Number of Major Thromboembolic Events Including Thrombotic Thrombocytopenic Purpura
Description: Major thromboembolic events (e.g., myocardial infarction, cerebrovascular accident, pulmonary embolism, or deep venous thrombosis) were assessed based on SMQ. Reported major thromboembolic events included TTP recurrences.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Number; unit: major thromboembolic events
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
major thromboembolic events | 11 | 4

10. Primary Outcome: Time to First Major Thromboembolic Event
Description: Time to first major thromboembolic event was defined as the duration of time (in days) from Baseline up to first major thromboembolic event in LTS16371. Participants without an event during LTS16371 were censored at the end of the study. Kaplan-Meier method was used for the analysis.
Time Frame: From Baseline up to 36 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
days | NA [845.00 to NA] — Median, upper limit of 95% CI were not calculated due to very few participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not calculated due to very few participants with events.

11. Primary Outcome: Cognitive Function: Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Total Absolute Scores at Baseline, 36 Months Follow-up Visit, and Change From Baseline in RBANS Total Score at 36 Months Follow-up Visit
Description: The RBANS is a 30-minute comprehensive screening test with five individual domains (immediate memory, delayed memory, attention, language, and visuospatial ability) to examine the cognitive mental status of a participant. Scores from all individual domain were aggregated into a total score and thus RBANS total score ranged from 40 to 160, where higher scores reflected better performance.
Time Frame: Baseline, 36 Months follow-up visit
Population: Analyzed on efficacy ITO population: participants who were enrolled in LTS16371 and did not experience aTTP recurrence in previous study ALX0681-C301 or prior to beginning of LTS16371. Here, 'number analyzed'=participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline: number analyzed (Participants) | 26 | 38
  Baseline | 89.7 (20.3) | 92.7 (14.9)
  At 36 Months: number analyzed (Participants) | 12 | 32
  At 36 Months | 98.0 (16.6) | 96.5 (17.0)
  Change at 36 Months: number analyzed (Participants) | 12 | 32
  Change at 36 Months | 2.1 (8.7) | 4.2 (8.9)

12. Primary Outcome: Health-Related Quality of Life (HRQoL): Change From Baseline in Headache Impact Test (HIT-6) Total Scores at Month 12, 24, and 36 Follow-up Visits
Description: HIT-6 is an easy to administer assessment that was used as a clinical evaluation of the impact of headache on a participant's QoL in both clinical practice and clinical research. The questionnaire included 6 questions covering the 6 areas of functioning most impacted in headache sufferers including pain, role functioning (the ability to carry out usual activities), social functioning, vitality (energy/ fatigue), cognitive functioning, and psychological/emotional distress. Total HIT-6 scores (sum of all individual questions) ranged from 36 (best outcome) to 78 (worst outcome), where higher scores indicated worse condition.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 45.0 (10.0) | 48.2 (9.9)
  Change at 12 Months: number analyzed (Participants) | 20 | 43
  Change at 12 Months | 0.9 (6.5) | 0.1 (7.0)
  Change at 24 Months: number analyzed (Participants) | 19 | 45
  Change at 24 Months | 1.2 (8.2) | -0.6 (8.7)
  Change at 36 Months: number analyzed (Participants) | 14 | 43
  Change at 36 Months | 0.6 (7.9) | 1.4 (7.5)

13. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire (SF-36) Health Survey - Physical Functioning Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Physical functioning domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in physical functioning domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 68.3 (28.9) | 74.1 (23.6)
  Change at 12 Months: number analyzed (Participants) | 20 | 46
  Change at 12 Months | 1.3 (16.8) | 1.5 (24.1)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | -0.8 (18.2) | 5.7 (19.3)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | 5.7 (17.4) | 6.2 (18.9)

14. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Role Functioning/Physical Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Role Functioning/Physical domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in role functioning/physical domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 60.1 (31.9) | 65.9 (30.6)
  Change at 12 Months: number analyzed (Participants) | 19 | 46
  Change at 12 Months | -5.3 (19.3) | 7.7 (35.4)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | 4.1 (24.1) | 7.1 (28.0)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | 5.8 (20.0) | 3.6 (28.6)

15. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Role Functioning/Emotional Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Role functioning/emotional domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in role functioning/emotional domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 75.3 (25.6) | 75.0 (29.4)
  Change at 12 Months: number analyzed (Participants) | 19 | 46
  Change at 12 Months | -13.2 (31.0) | 1.6 (38.0)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | -1.3 (32.5) | 0.9 (33.7)
  Change at 36 Month: number analyzed (Participants) | 15 | 43
  Change at 36 Month | -4.4 (20.6) | -3.7 (29.6)

16. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Energy/Fatigue Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Energy/fatigue domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in energy/fatigue domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 50.9 (21.2) | 52.4 (20.9)
  Change at 12 Months: number analyzed (Participants) | 20 | 45
  Change at 12 Months | -0.3 (18.3) | 2.0 (20.7)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | 5.9 (21.4) | 0.6 (21.7)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | 7.5 (21.3) | 3.9 (18.7)

17. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Emotional Well-being Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Emotional well-being domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in emotional well-being domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 72.1 (18.3) | 70.1 (20.7)
  Change at 12 Months: number analyzed (Participants) | 20 | 45
  Change at 12 Months | -9.3 (18.2) | -2.5 (21.1)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | -3.3 (18.9) | -2.0 (21.3)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | -0.7 (14.6) | -1.5 (19.3)

18. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Social Functioning Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Social functioning domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in social functioning domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 74.6 (25.3) | 74.0 (28.5)
  Change at 12 Months: number analyzed (Participants) | 20 | 46
  Change at 12 Months | -10.6 (26.7) | 1.6 (35.1)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | 0.0 (27.5) | -0.8 (33.8)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | 0.8 (18.0) | -2.6 (31.9)

19. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Pain Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Pain domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in pain domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 68.4 (31.7) | 68.0 (23.5)
  Change at 12 Months: number analyzed (Participants) | 20 | 46
  Change at 12 Months | -1.8 (30.4) | 0.3 (33.6)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | -9.4 (32.5) | 5.0 (24.9)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | -5.2 (21.5) | 3.7 (25.6)

20. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - General Health Domain Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. General Health domain scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in general health domain score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 66.4 (18.5) | 53.1 (19.3)
  Change at 12 Months: number analyzed (Participants) | 20 | 46
  Change at 12 Months | -4.0 (19.8) | 4.9 (19.0)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | -1.5 (17.9) | 4.8 (20.9)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | -4.7 (11.1) | 3.6 (17.3)

21. Primary Outcome: Health-Related Quality of Life: Change From Baseline in 36-Item Short Form Questionnaire Health Survey - Change in Health Status Scores at Month 12, 24, and 36 Follow-up Visits
Description: The SF-36 consisted of 36 items that was summarized into 8 domains: physical functioning, social functioning, role functioning/physical, role functioning/emotional, emotional well-being, energy/fatigue, pain, general health and an additional single item covering change in health status. Change in health status scores ranged from 0 (worst value) to 100 (best value), with higher scores reflecting better health status. Change from baseline in change in health status score at months 12, 24, and 36 were reported in this outcome measure.
Time Frame: Baseline, Month 12, 24, and 36 Follow-up visits
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 49
units on a scale
  Baseline | 45.7 (31.4) | 53.6 (34.2)
  Change at 12 Months: number analyzed (Participants) | 20 | 46
  Change at 12 Months | 30.0 (40.2) | 20.1 (44.0)
  Change at 24 Months: number analyzed (Participants) | 20 | 45
  Change at 24 Months | 21.3 (36.5) | 10.6 (39.0)
  Change at 36 Months: number analyzed (Participants) | 15 | 43
  Change at 36 Months | 16.7 (33.6) | 4.7 (37.1)

22. Primary Outcome: Percentage of Participants With Drug-induced Treatment-emergent (TE) Anti-drug Antibodies (ADA) Positive Response
Description: Drug-induced TE ADA positive was based on the outcome of a tiered assay approach that included a modified ADA (mADA) method to eliminate the effects of pre-existing antibodies (pre-Ab). TE ADA responses reported here included both pre-Ab positive and negative responses. A participant was considered as drug-induced TE ADA positive if post-dose samples were positive, regardless of the status of pre-dose samples in the ADA and modified ADA assay.
Time Frame: From Baseline up to 36 months
Population: Analysis was performed on overall ITO population which included participants who were enrolled in LTS16371, grouped by whether they received caplacizumab during previous study ALX0681-C301 versus those who never received caplacizumab before enrollment in LTS16371.
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 75
percentage of participants | 0 | 10.7

23. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with the treatment. An SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event.
Time Frame: From Baseline up to 36 months
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
Number analyzed (Participants) | 29 | 75
Participants
  At least one AE | 26 | 68
  At least one SAE | 16 | 28
  At least one AE leading to death | 1 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to 36 months
Description: Analysis was performed on overall ITO population which included participants who were enrolled in LTS16371, grouped by whether they received caplacizumab during previous study ALX0681-C301 versus those who never received caplacizumab before enrollment in LTS16371.
Arm/Group | Standard of Care (SoC) (Treated in Study C301) | Caplacizumab (Treated in Study C301)
All-Cause Mortality (participants affected / at risk) | 1/29 | 0/75
Serious Adverse Events (participants affected / at risk) | 16/29 | 28/75
Other Adverse Events (participants affected / at risk) | 22/29 | 58/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (Treated in Study C301) (N=29) | Caplacizumab (Treated in Study C301) (N=75)
Allergic Transfusion Reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (3) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 8 (9) | 11 (21)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glomerulonephritis Membranous (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage Urinary Tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Infarct (Renal and urinary disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis Viral (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Meningitis Aseptic (Infections and infestations) | 0 (0) | 1 (1)
Ophthalmic Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (3)
Pneumonia Pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Abortion Induced (Surgical and medical procedures) | 0 (0) | 2 (2)
Cholecystectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hysterocele (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (Treated in Study C301) (N=29) | Caplacizumab (Treated in Study C301) (N=75)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Adamts13 Activity Decreased (Investigations) | 0 (0) | 13 (13)
Blood Cholesterol Increased (Investigations) | 0 (0) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 10 (10)
Headache (Nervous system disorders) | 9 (9) | 16 (17)
Paraesthesia (Nervous system disorders) | 5 (5) | 4 (4)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Iron Deficiency (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Bronchitis (Infections and infestations) | 0 (0) | 5 (5)
Herpes Zoster (Infections and infestations) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 7 (7)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 4 (4)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1)
Tooth Abscess (Infections and infestations) | 2 (2) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 4 (5)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 2 (2) | 4 (5)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 7 (7)
Pyrexia (General disorders) | 3 (3) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02878603/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT02878603/SAP_001.pdf